CLINICAL TRIAL: NCT01742377
Title: i-Scan Endoscopy in the Detection of Minimal Change Esophagitis in Dyspeptic Patients With or Without Gastroesophageal Reflux Disease by Gerd Q Questionnaire and by 24 Hour pH Monitoring.
Brief Title: Minimal Change Esophagitis by i-Scan Endoscopy in Dyspeptic Patients
Acronym: MCE
Status: Completed | Type: Observational
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Nisa Netinatsunton, NKC Institute of Gastrornterology and Hepatology, Prince of Songkla University
Other Study IDs: EC 53-017-21-1-2
Record Dates: First submitted 2012-10-28; First posted 2012-12-05 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-01

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD; Dyspepsia; Ambulatory 24-hour Esophageal pH Monitoring; Minimal change erosions
MeSH Terms: conditions — Gastroesophageal Reflux; Dyspepsia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Patients with GerdQ positive: Gerd Q positive was defined as score equal or more than eight.
  Interventions: Procedure: Patients with GerdQ positive
- Patients with GerdQ negative: Gerd Q neegative was defined as score less than eight.
  Interventions: Procedure: Patients with GerdQ negative
- Normal volunteers: Normal volunteers was defined as population without dyspeptic symptom.
  Interventions: Procedure: Normal volunteers

INTERVENTIONS:
Procedure: Patients with GerdQ positive — Patients done GerdQ questionnaire, then undergone EGD. The distal esophagus was examined by HD and followed by SE with a preset TE mode for esophagus ( TE-e mode ). All patients had pH monitoring study within 1 week after the endoscopy.
  Groups: Patients with GerdQ positive
Procedure: Patients with GerdQ negative — Patients done GerdQ questionnaire, then undergone EGD. The distal esophagus was examined by HD and followed by SE with a preset TE mode for esophagus ( TE-e mode ). All patients had pH monitoring study within 1 week after the endoscopy.
  Groups: Patients with GerdQ negative
Procedure: Normal volunteers — Normal volunteers undergone EGD.The distal esophagus was examined by HD and followed by SE with a preset TE mode for esophagus ( TE-e mode ).
  Groups: Normal volunteers

SUMMARY:
The purpose of this study to assess efficacy of SE endoscopy in the detection of MCE in dyspeptic patients with or without GERD diagnosed by GerdQ or by endoscopy + PHM and in normal volunteers.

DETAILED DESCRIPTION:
Background: The association of minimal change esophagitis (MCE) with gastroesophageal reflux (GERD) is controversy. High resolution endoscopy may improve the detection of minimal change lesion (MCL). i- Scan endoscopy (SE) provides high resolution images with modulation of images for a specific purpose.

Methods. All dyspeptic patients with or without GERD symptoms scheduled for endoscopy were recruited from February 2010 till July 2014. All completed the validated Thai version of GerdQ then underwent endoscopy. Forty normal volunteers were recruited for endoscopy and PHM test. The esophagus was examined by HD and SE with the TE-e mode sequentially. The captured images were independently evaluated for MCL (punctate erythema (PE), minute erosion (ME) and triangular lesion with elongated pit (EP) by three endoscopists. The agreement of > 2 endoscopists was accepted as a final result. All had PHM within 1 week after the endoscopy. GERD was diagnosed by LA grade A-D esophagitis and/or PHM with acid exposure time > the upper limit of volunteer and/or positive symptom index and/or positive Symptom Association Probability. MCE was diagnosed when PE, ME or EP or the combination of these were present.

The 40 normal volunteers were recruited for performing pH monitoring. The PHM data of 40 volunteers were analyzed to set the upper normal limit of total acid exposure time in our population. The mean + 2SD of total acid exposure time of volunteers was 1.9%.

Definition. GerdQ. The Thai version of GerdQ was translated from the English version. The contents of the GerdQ were tested by back translation from Thai to English by 5 personnel who are fluent in English and all showed the consistent contents. The reliability of the GerdQ was validated in 22 volunteers completing the questionnaire twice with 3 hours in between and showed no significant difference of the mean score (5.14+ 2.34 vs 6.23+ 1.57, p=0.07) and the number of subjects with GERD diagnosed by the GerdQ (2 vs 5, Fisher's extact test, p=0.21) .

GERD is diagnosed when total acid exposure time is more than 2% or positive symptom index (SI) or positive symptom association probability ( SAP ) or endoscopy revealed LA erosive esophagitis > grade A.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one or more of the following symptoms namely epigastric pain or discomfort, postprandial fullness and early satiety with or without symptoms suggesting GERD
* Patients able to give informed consent

Exclusion Criteria:

* Patients with significant weight loss.
* Patients with hematemesis, melena ,dysphagia, intractable vomiting , palpable abdominal mass.
* Patients with history of documented peptic ulcer , gastric surgery , gastric cancer.
* Patients with symptoms compatible with irritable bowel syndrome, hepatobiliary tract disease.
* Patients with severe concomitant medical conditions, pregnant woman or continuous usage of steroids or NSIADS in the preceding 1 month before entry to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with dyspepsia from clinics , primary care clinics ,community.
Sampling Method: Non-Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2010-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Evidence of minimal change erosions detected by i-scan endoscopy. | within day of endoscopy
  Minimal change lesions (MCL) included punctate erythema (PE), minute erosion (ME) and triangular lesion with elongated pit (TLE).

SECONDARY OUTCOMES:
Number of patients with dyspepsia are diagnosed gastroesophageal reflux disease by Gerd Q. | within the first 7 days after endoscopy
  The GerdQ score equal or more than 8 is a positive score for GERD
Number of patients with dyspepsia are confirmed with GERD | within the first 7 days after endoscopy
  GERD is diagnosed when total acid exposure time is more than 2% or positive symptom index (SI) or positive symptom association probability ( SAP ) or endoscopy revealed LA erosive esophagitis > grade A .
Total acid exposure in normal volunteers | 1 day
  The mean value of total acid exposure of 40 normal volunteer.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Nisa Netinatsunton, MD, Principal Investigator — NKC Institue of Gastroenterology and Hepatology,Prince of Songkla University
Locations (1):
- NKC Institue of Gastroenterology and Hepatology, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

REFERENCES:
- [Derived] Netinatsunton N, Sottisuporn J, Attasaranya S, Witeerungrot T, Chamroonkul N, Jongboonyanuparp T, Geater A, Ovartlarnporn B. i-Scan detection of minimal change esophagitis in dyspeptic patients with or without Gastroesophageal Reflux disease. BMC Gastroenterol. 2016 Jan 14;16:4. doi: 10.1186/s12876-016-0417-4. PMID 26762316